CLINICAL TRIAL: NCT02697227
Title: Low Reward Sensitivity and Behavioral Activation Therapy for Smoking Cessation
Brief Title: Behavioral Activation Therapy and Nicotine Replacement Therapy in Increasing Smoking Cessation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2015-0879; NCI-2016-00674 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0879 (Other: M D Anderson Cancer Center); R34DA037391 (NIH)
Record Dates: First submitted 2016-02-24; First posted 2016-03-03 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Cigarette Smoker; Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Behavior Therapy; Tobacco Use Cessation Devices; Nicotine; Smoking Devices

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Group I (NRT, SC) (Active Comparator): Patients receive NRT patch daily for 8 weeks. Patients receive individual behavioral treatment sessions consisting of behavioral treatment strategies for smoking cessation and health education information over 45 minutes for 8 sessions.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Nicotine Patch; Other: Questionnaire Administration; Behavioral: Smoking Cessation Intervention
- Group II (NRT, BATS) (Active Comparator): Patients receive NRT patch daily for 8 weeks. Patients complete individual treatment sessions consisting of SC strategies and BA strategies over 45 minutes for 8 sessions.
  Interventions: Behavioral: Behavioral Intervention; Other: Laboratory Biomarker Analysis; Drug: Nicotine Patch; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Receive BATS counseling
  Other Names: Behavior Conditioning Therapy; behavior modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; BEHAVIORAL THERAPY; Behavioral Treatment; Behavioral Treatments
  Arms: Group II (NRT, BATS)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nicotine Patch — Receive nicotine patch
  Other Names: NicoDerm CQ; Nicotine Skin Patch; Nicotine Transdermal Patch
Other: Questionnaire Administration — Ancillary studies
Behavioral: Smoking Cessation Intervention — Receive standard smoking cessation counseling
  Other Names: Smoking and Tobacco Use Cessation Interventions
  Arms: Group I (NRT, SC)

SUMMARY:
This randomized clinical trial studies how well behavioral activation therapy and nicotine replacement therapy work in increasing smoking cessation. Behavioral interventions use techniques to help patients change the way they react to environmental triggers that may cause a negative reaction. Giving behavioral activation therapy and nicotine replacement therapy may help patients quit smoking or change their smoking behavior.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the comparative effectiveness of Behavioral Activation Treatment for Smoking (BATS) plus nicotine replacement therapy (NRT) versus standard cessation treatment plus NRT on high reward sensitivity smokers (IRS+) and low reward sensitivity (IRS-) smokers.

II. To identify mediators of the BATS plus NRT treatment effect in IRS- smokers.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I (STANDARD CESSATION): Patients receive NRT patch daily for 8 weeks. Patients receive individual behavioral treatment sessions consisting of behavioral treatment strategies for smoking cessation and health education information over 45 minutes for 8 sessions.

GROUP II (BATS): Patients receive NRT patch daily for 8 weeks. Patients receive individual treatment sessions consisting of standard cessation (SC) strategies and behavioral activation (BA) strategies over 45 minutes for 8 sessions.

After completion of study intervention, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Smoking 5 or more cigarettes, little cigars or cigarillos per day, on average, within the 2 months preceding the screening visit and expired carbon monoxide (CO) greater than or equal to 6 parts per million (ppm); (if < 6, then NicAlert Strip > 2)
* Interested in treatment that might change smoking behavior
* Able to follow verbal and written instructions in English and complete all aspects of the study
* Provide informed consent and agree to all assessments and study procedures
* Have an address and telephone number where they may be reached
* Be the only participant in their household

Exclusion Criteria:

* Within the month immediately preceding the screening visit, use of any form of tobacco products other than cigarettes, little cigars or cigarillos on 3 or more days within a week if the individual refuses to refrain from such tobacco use during the course of the study
* Current enrollment or plans to enroll in another smoking cessation program in the next 6 months
* Plan to use other nicotine substitutes (i.e., over-the-counter [OTC] or prescription medication for smoking cessation) or smoking cessation treatments in the next 6 months
* Uncontrolled hypertension (systolic blood pressure [SBP] greater than 180 or diastolic blood pressure [DBP] greater than 110)
* Reports diagnosis of seizure disorder or a history of neurological illness or closed head injury that in the opinion of the principal investigator (PI) or designated expert(s) feels that it would affect the results of the electroencephalogram (EEG)
* Current use of certain medications:

  * Smoking cessation meds (last 7 days), i.e., Wellbutrin, bupropion, Zyban, NRT, Chantix
  * Certain medications to treat depression (last 14 days), i.e. monoamine oxidase inhibitors (MAOIs) and Elavil (amitriptyline), or
  * Other medications listed on the exclusionary medications list
* Meet criteria for the following psychiatric and/or substance use disorders as assessed by the Mini International Neuropsychiatric Interview (MINI): items C (current manic or hypomanic episode only), I (alcohol abuse - alcohol addendum-past 6 months only; current alcohol dependence), J (substance abuse - substance abuse addendum - past 6 months only; current substance dependence), K (psychotic disorder or mood disorder with psychotic features); individuals who meet criteria for non-exclusionary psychiatric disorders that are considered clinically unstable and/or unsuitable to participate as determined by the principal investigator
* Individuals rated as moderate (9-16) to high (17 or greater) on suicidality as assessed by module B of the MINI
* Psychiatric hospitalization within 1 year of screening date
* A positive urine pregnancy test during the screening period; women who are two years post-menopausal, or who have had a tubal ligation or a partial or full hysterectomy will not be subject to a urine pregnancy test
* Pregnant, breast-feeding or of childbearing potential and is not protected by a medically acceptable, effective method of birth control while enrolled in the study; medically acceptable contraceptives include: (1) approved hormonal contraceptives (such as birth control pills, patches, implants or injections), (2) barrier methods (such as a condom or diaphragm) used with a spermicide, or (3) an intrauterine device (IUD); contraceptive measures sold for emergency use after unprotected sex are not acceptable methods for routine use
* History of hypersensitivity or allergic reaction to NRT, or any component of its formulation
* Any medical or psychiatric condition, illness, disorder, or concomitant medication that could compromise participant safety or treatment, as determined by the principal investigator
* Subject considered by the investigator as unsuitable candidate for receipt of NRT, or unstable to be followed up throughout the entire duration of the study
* Must not have visual problems that in the investigators opinion would interfere in the completion of the study assessments
* Unwilling to change hairstyle or remove a wig as necessary for the appointment to accommodate the net that is required to be worn on the scalp during the study procedure
* Positive toxicology screen for any of the following drugs: cocaine, opiates, methadone, benzodiazepines, barbiturates, amphetamines, methamphetamines, or phencyclidine (PCP)

  * Participants with valid prescriptions for opiates, benzodiazepines, barbiturates, amphetamines or methadone will not be excluded
  * Participants failing the toxicology screen will be allowed to re-screen once; if they test positive again, they will not be allowed to return for 90 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2016-08-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of behavioral activation treatment for smoking plus nicotine replacement therapy versus standard cessation treatment plus nicotine replacement therapy defined as abstinence rate in low reward sensitivity- and + smokers | Up to 4 months
Mediators of the behavioral activation treatment for smoking plus nicotine replacement therapy treatment effect in low reward sensitivity- smokers | Up to 4 months
  The primary outcome measure is cigarettes per day (CPD) as measured by Time Line Follow Back. This self-report will be biochemically verified by either carbon monoxide breath sample or nicotine sample

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Minnix, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org